CLINICAL TRIAL: NCT03114137
Title: Heart, Arteries and Sikle Cell Disease, a Multicentric Cohort of Cardiovascular Complications in Subsaharan Africa
Brief Title: Heart Arteries and Sickle Cell Disease / Coeur Artères DREpanocytose
Acronym: CADRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiologie et Développement (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Paris 5 - Rene Descartes (Other); laboratory of excellence GR-Ex (Unknown)
Responsible Party: Principal Investigator, Xavier Jouven, Professor, Cardiologie et Développement
Other Study IDs: 002
Record Dates: First submitted 2017-03-30; First posted 2017-04-14 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Sickle Cell Anemia; Sickle Cell Disease
Keywords: Sub-Saharan Africa; Sickle Cell Disease; Vasculopathy; Nephropathy; Pulmonary hypertension; cardiac disease; hemolysis; pulse wave velocity; blood viscosity
MeSH Terms: conditions — Anemia, Sickle Cell; Vascular Diseases; Kidney Diseases; Hypertension, Pulmonary; Heart Diseases; Hemolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood plasma saliva urines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sickle cell patients: * age: five-year-old or more
  * major sickle cell syndrome confirmed by hemoglobin phenotype: SS, SC, SBeta+ or Sbeta0
  * steady state defined as the absence of vaso-occlusive crisis for the previous 15 days, absence of fever or infectious disease for the previous 8 days and absence of transfusion for the previous 2 months
- control patients: * volunteer parents or siblings of sickle cell patients
  * hospital staff or their children matched on country and age +/- 3 ans with the patients

SUMMARY:
The CADRE study is a multinational observational cohort of patients with sickle-cell disease (SCD) in five west and central sub-Saharan African countries. The aim of this project is to describe the incidence and assess the predictive factors of SCD-related micro- and macro-vascular complications in sub-Saharan Africa.

DETAILED DESCRIPTION:
Sickle cell disease (SCD), one of the lost common genetic diseases worldwide, is caused by a mutation in the β globin gene. Most patients with this disease are homozygous for the βS allele (SS), whereas others have inherited a βS allele with another mutation in the β globin gene. In addition to repeated acute ischemic insults due to the red blood cells sickling in the microcirculation, a chronic vasculopathy leads to organ injuries, such as kidney disease, stroke, pulmonary hypertension, retinopathy, bone infarcts, and leg ulcers.

CADRE is a multinational prospective observational study undertaken in five countries in sub-Saharan Africa. Patients with SCD will be recruited through outpatients' clinics in public, university and private hospitals and research centers in five countries. The CADRE protocol was approved by the relevant national ethics committee in each of the participating countries.

Primary endpoint is to measure the prevalence and the incidence of the main vascular complications in the main types of SCD: glomerulopathy, nephropathy, cardiopathy, pulmonary hypertension, retinopathy, strokes, osteonecrosis and leg ulcers.

Secondary endpoints are:

* to define the clinical and biological predictors of SCD vasculopathy in Africa
* to search for genetic risk factors for the SCD-related cardiovascular complications, in particular alpha thalassemia, persistence of foetal hemoglobin and other candidate genetic polymorphisms
* to search for functional risk factors (pulse wave velocity, capillary vasodilatation, blood visosity) for the SCD-related cardiovascular complications
* to search for new biological determinant of SCD-related cardiovascular complications, in particular alternative markers of hemolysis (microparticules, free heme) and inflammation (cytokines, leucocytes phenotyping, NET (neutrophile extracellular traps))

ELIGIBILITY:
Inclusion Criteria:

* age: five-year-old or more
* signature of informed consent Patients : major sickle cell syndrome confirmed by hemoglobin phenotyping: SS, SC, SBeta+ or Sbeta0 Controls : healthy parents or siblings of the patients, hospital staff or their children, matched on age+/- 3 years and country (1 control for 4 patients)

Exclusion Criteria:

unstable clinical status such as:

* vaso-occlusive crisis in the previous 15 days
* fever or infectious disease in the previous 15 days
* transfusion in the previous 2 months

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adult patients with the sickle cell disease living in subSaharan Africa
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence and 10 year-incidence of SCD-related vascular complications in different phenotypes of SCD: glomerulopathy | 10 years
  urinary albumin/creatinin ratio (mg/g)
Prevalence and 10 year-incidence of SCD-related vascular complications in different phenotypes of SCD: cardiopathy | 10 years
  left ventricular ejection fraction < 60 %
Prevalence and 10 year-incidence of SCD-related vascular complications in different phenotypes of SCD: pulmonary hypertension | 10 years
  tricuspid regurgitation jet velocity (m/s)
Prevalence and incidence and the 10 year-incidence of the main SCD-related vascular complications in different phenotypes of SCD: retinopathy | 10 years
  retinal examination
Prevalence and 10 year-incidence of SCD-related vascular complications in different phenotypes of SCD:stroke | 10 years
  clinical diagnosis
Prevalence and 10 year-incidence of SCD-related vascular complications in different phenotypes of SCD:osteonecrosis | 10 years
  standard radiography
Prevalence and 10 year-incidence of SCD-related vascular complications in different phenotypes of SCD: leg ulcers | 10 years
  clinical diagnosis
Prevalence and 10 year-incidence of SCD-related vascular complications in different phenotypes of SCD: priapism | 10 years
  clinical diagnosis

SECONDARY OUTCOMES:
Potential biological risk marker measured at baseline and follow up visits: carotid-femoral pulse wave velocity | 10 years
  measured by Pulsepen, m/s)
Potential biological risk marker measured at baseline and follow up visits: complete blood count | 10 years
Potential biological risk marker measured at baseline and follow up visits: LDH level | 10 years
Potential biological risk marker measured at baseline and follow up visits: bilirubin level | 10 years
Potential biological risk marker measured at baseline and follow up visits: microparticules measure | 10 years
Potential biological risk marker measured at baseline and follow up visits: free heme level | 10 years
Potential biological risk marker measured at baseline and follow up visits: inflammatory cytokines | 10 years
Potential biological risk marker measured at baseline and follow up visits: neutrophil extracellular traps | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Jouven, MD PhD, Principal Investigator — Cardiologie et Developpement
Locations (13):
- Cameroon (4):
  - Central Hospital of Yaounde, Yaoundé
  - Centre mère et enfant / fondation Chantal Biya, Yaoundé
  - Centre Pasteur du Cameroun, Yaoundé
  - Pediatrics unit, Centre Hospitalier d'Essos, Yaoundé
- Côte d’Ivoire (2):
  - Hematology Unit, CHU Yopougon, Abidjan
  - Institut de cardiologie, Abidjan
- Centre hospitalier Monkole, Kinshasa, Democratic Republic of the Congo
- CIRMF, Libreville, Gabon
- Mali (2):
  - Cardiology Unit, Centre gyneco-obstretrique, Bamako
  - Centre de Recherche et de Lutte contre la Drepanocytose, Bamako
- Senegal (3):
  - Centre hospitalier d'enfants Albert Royer, Dakar
  - Centre hospitalo-universotaire de Fann, Cardiology department, Dakar
  - Centre national de transfusion sanguine, Dakar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kato GJ, Gladwin MT, Steinberg MH. Deconstructing sickle cell disease: reappraisal of the role of hemolysis in the development of clinical subphenotypes. Blood Rev. 2007 Jan;21(1):37-47. doi: 10.1016/j.blre.2006.07.001. Epub 2006 Nov 7. PMID 17084951
- [Background] Hebbel RP. Reconstructing sickle cell disease: a data-based analysis of the "hyperhemolysis paradigm" for pulmonary hypertension from the perspective of evidence-based medicine. Am J Hematol. 2011 Feb;86(2):123-54. doi: 10.1002/ajh.21952. PMID 21264896
- [Background] Nouraie M, Lee JS, Zhang Y, Kanias T, Zhao X, Xiong Z, Oriss TB, Zeng Q, Kato GJ, Gibbs JS, Hildesheim ME, Sachdev V, Barst RJ, Machado RF, Hassell KL, Little JA, Schraufnagel DE, Krishnamurti L, Novelli E, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Castro OL, Goldsmith JC, Gordeuk VR, Gladwin MT; Walk-PHASST Investigators and Patients. The relationship between the severity of hemolysis, clinical manifestations and risk of death in 415 patients with sickle cell anemia in the US and Europe. Haematologica. 2013 Mar;98(3):464-72. doi: 10.3324/haematol.2012.068965. Epub 2012 Sep 14. PMID 22983573
- [Background] Gordeuk VR, Minniti CP, Nouraie M, Campbell AD, Rana SR, Luchtman-Jones L, Sable C, Dham N, Ensing G, Prchal JT, Kato GJ, Gladwin MT, Castro OL. Elevated tricuspid regurgitation velocity and decline in exercise capacity over 22 months of follow up in children and adolescents with sickle cell anemia. Haematologica. 2011 Jan;96(1):33-40. doi: 10.3324/haematol.2010.030767. Epub 2010 Sep 30. PMID 20884713
- [Background] Maier-Redelsperger M, Levy P, Lionnet F, Stankovic K, Haymann JP, Lefevre G, Avellino V, Perol JP, Girot R, Elion J. Strong association between a new marker of hemolysis and glomerulopathy in sickle cell anemia. Blood Cells Mol Dis. 2010 Dec 15;45(4):289-92. doi: 10.1016/j.bcmd.2010.08.001. Epub 2010 Sep 15. PMID 20833087
- [Background] Taylor JG 6th, Nolan VG, Mendelsohn L, Kato GJ, Gladwin MT, Steinberg MH. Chronic hyper-hemolysis in sickle cell anemia: association of vascular complications and mortality with less frequent vasoocclusive pain. PLoS One. 2008 May 7;3(5):e2095. doi: 10.1371/journal.pone.0002095. PMID 18461136
- [Background] Gladwin MT, Sachdev V, Jison ML, Shizukuda Y, Plehn JF, Minter K, Brown B, Coles WA, Nichols JS, Ernst I, Hunter LA, Blackwelder WC, Schechter AN, Rodgers GP, Castro O, Ognibene FP. Pulmonary hypertension as a risk factor for death in patients with sickle cell disease. N Engl J Med. 2004 Feb 26;350(9):886-95. doi: 10.1056/NEJMoa035477. PMID 14985486
- [Background] Kato GJ, McGowan V, Machado RF, Little JA, Taylor J 6th, Morris CR, Nichols JS, Wang X, Poljakovic M, Morris SM Jr, Gladwin MT. Lactate dehydrogenase as a biomarker of hemolysis-associated nitric oxide resistance, priapism, leg ulceration, pulmonary hypertension, and death in patients with sickle cell disease. Blood. 2006 Mar 15;107(6):2279-85. doi: 10.1182/blood-2005-06-2373. Epub 2005 Nov 15. PMID 16291595
- [Background] Connes P, Lamarre Y, Hardy-Dessources MD, Lemonne N, Waltz X, Mougenel D, Mukisi-Mukaza M, Lalanne-Mistrih ML, Tarer V, Tressieres B, Etienne-Julan M, Romana M. Decreased hematocrit-to-viscosity ratio and increased lactate dehydrogenase level in patients with sickle cell anemia and recurrent leg ulcers. PLoS One. 2013 Nov 4;8(11):e79680. doi: 10.1371/journal.pone.0079680. eCollection 2013. PMID 24223994
- [Background] Nolan VG, Wyszynski DF, Farrer LA, Steinberg MH. Hemolysis-associated priapism in sickle cell disease. Blood. 2005 Nov 1;106(9):3264-7. doi: 10.1182/blood-2005-04-1594. Epub 2005 Jun 28. PMID 15985542
- [Background] Kato GJ, Hsieh M, Machado R, Taylor J 6th, Little J, Butman JA, Lehky T, Tisdale J, Gladwin MT. Cerebrovascular disease associated with sickle cell pulmonary hypertension. Am J Hematol. 2006 Jul;81(7):503-10. doi: 10.1002/ajh.20642. PMID 16755569
- [Background] Steinberg MH, Sebastiani P. Genetic modifiers of sickle cell disease. Am J Hematol. 2012 Aug;87(8):795-803. doi: 10.1002/ajh.23232. Epub 2012 May 28. PMID 22641398
- [Result] Ranque B, Menet A, Boutouyrie P, Diop IB, Kingue S, Diarra M, N'Guetta R, Diallo D, Diop S, Diagne I, Sanogo I, Tolo A, Chelo D, Wamba G, Gonzalez JP, Abough'elie C, Diakite CO, Traore Y, Legueun G, Deme-Ly I, Faye BF, Seck M, Kouakou B, Kamara I, Le Jeune S, Jouven X. Arterial Stiffness Impairment in Sickle Cell Disease Associated With Chronic Vascular Complications: The Multinational African CADRE Study. Circulation. 2016 Sep 27;134(13):923-33. doi: 10.1161/CIRCULATIONAHA.115.021015. Epub 2016 Aug 31. PMID 27582423
- [Result] Ranque B, Menet A, Diop IB, Thiam MM, Diallo D, Diop S, Diagne I, Sanogo I, Kingue S, Chelo D, Wamba G, Diarra M, Anzouan JB, N'Guetta R, Diakite CO, Traore Y, Legueun G, Deme-Ly I, Belinga S, Boidy K, Kamara I, Tharaux PL, Jouven X. Early renal damage in patients with sickle cell disease in sub-Saharan Africa: a multinational, prospective, cross-sectional study. Lancet Haematol. 2014 Nov;1(2):e64-73. doi: 10.1016/S2352-3026(14)00007-6. Epub 2014 Oct 28. PMID 27030156
- [Derived] Ranque B, Diaw M, Dembele AK, Lapoumeroulie C, Offredo L, Tessougue O, Gueye SM, Diallo D, Diop S, Colin-Aronovicz Y, Jouven X, Blanc-Brude O, Tharaux PL, Le Jeune S, Connes P, Romana M, Le Van Kim C. Association of haemolysis markers, blood viscosity and microcirculation function with organ damage in sickle cell disease in sub-Saharan Africa (the BIOCADRE study). Br J Haematol. 2023 Oct;203(2):319-326. doi: 10.1111/bjh.19006. Epub 2023 Aug 15. PMID 37583261
- [Derived] Dembele AK, Lapoumeroulie C, Diaw M, Tessougue O, Offredo L, Diallo DA, Diop S, Elion J, Colin-Aronovicz Y, Tharaux PL, Jouven X, Romana M, Ranque B, Le Van Kim C. Cell-derived microparticles and sickle cell disease chronic vasculopathy in sub-Saharan Africa: A multinational study. Br J Haematol. 2021 Feb;192(3):634-642. doi: 10.1111/bjh.17242. Epub 2020 Nov 29. PMID 33249569